CLINICAL TRIAL: NCT01762111
Title: AMH and Pregnancy Rate by Age During Stimulate In-Vitro Fertilization Protocol
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: OVO-12-22
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility
Keywords: Anti-Mullerian Hormone; In-Vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The woman fertility decrease with the age and there is a closely link with the ovarian reserve, the number of available eggs in the ovaries. Therefore, it is important to evaluate the ovarian reserve with specific marker to have a better prediction of the response of the in vitro fertilization treatment and to have a better rate of pregnancy.

Until now, a lot of clinical criteria (age, duration of the infertility, number of antral follicles) and biological (FSH, Oestradiol, Inhibin B, EFFORT test, number of the eggs at the retrieval day) was suggested to help for the estimation of the ovarian reserve.

Since couple of years, the anti-müllerian hormone (AMH) is recognize to be one of the best ovarian reserve marker, it corresponding the number of antral follicles, it is more sensitive and predictive. Moreover, during the In-Vitro Fertilization, the anti-müllerian hormone can provide the weak responds at the stimulation and the reverse, the risk of excessive responds (hyperstimulation). To choose the gonadotropin doses to administrate (stimulation ovarian hormone) during an In-Vitro Fertilization protocol, we need to know the anti-müllerian hormone dosage. However, if the anti-müllerian hormone is recognize to evaluate the quantity of available eggs in the ovaries, his role to determine the quality of these eggs still discussed.

The goal of this study is to verify if the serum anti-müllerian hormone (blood) is a good indicator for the quality of the reserve ovarian evaluating the impact of anti-müllerian hormone rate on the pregnancy rate and implantation rate, during stimulate In-Vitro Fertilization protocol.

ELIGIBILITY:
Inclusion Criteria:

* All infertile patients aged between 18 and 43 years
* Patients with a prescription for a stimulated In-Vitro Fertilization cycle

Exclusion Criteria:

* Presence of endocrine disease: diabetes, hyperprolactinemia, abnormal thyroid-stimulating hormone (TSH) or Cushing syndrome
* Renal or hepatic impairment known

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women followed at the clinique ovo, aged between 18 and 43 years old undergoing a stimulate In-Vitro Fertilization cycle.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates | 7 weeks
  Clinical pregnancy rates per cycle and per transfer

SECONDARY OUTCOMES:
Cumulative pregnancy rates | 5 years
  Cumulative pregnancy rates including all frozen embryo transfer
Number of eggs | 4 weeks
  Number of eggs retrieve at the end of the stimulated in-vitro fertilization cycle
Number of embryos | 4 weeks
  Number of embryos obtain at the end of the stimulated in-vitro fertilization cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada